CLINICAL TRIAL: NCT00580359
Title: A Randomized Phase II Study of S-1 Versus Capecitabine as First-Line Chemotherapy in the Elderly and/or Poor Performance Status Patients With Recurrent or Metastatic Gastric Cancer
Brief Title: S-1 vs Capecitabine in the Elderly and/or Poor Performance Status Patients With Recurrent or Metastatic Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Sook Ryun Park, M.D., National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-07-263
Record Dates: First submitted 2007-12-21; First posted 2007-12-24 (Estimated); Last update posted 2008-01-08 (Estimated); Status verified 2007-12

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms; Secondary; Combination chemotherapy; S-1; Capecitabine
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — S 1 (combination); Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): S-1 40mg/m2 orally twice daily on days 1 (evening) - 15 (morning)
  Interventions: Drug: S-1, capecitabine
- B (Active Comparator): Capecitabine 1250mg/m2 orally twice daily on days 1 (evening) - 15 (morning)
  Interventions: Drug: S-1, capecitabine

INTERVENTIONS:
Drug: S-1, capecitabine — S-1 40mg/m2 orally twice daily on days 1(evening) - 15 (morning)every 3 weeks, until disease progression, Capecitabine 1250mg/m2 orally twice daily on days 1 (evening) - 15 (morning)every 3 weeks, until disease progression

SUMMARY:
This study is an open-label, single-center, and randomized phase II study designed to evaluate each efficacy and safety of S-1 and capecitabine in the elderly and/or poor performance status patients with recurrent or metastatic gastric cancer. The randomization will be stratified by age (70-85 years versus 65 years and < 70 years) and performance status, which is dependent on age group; in 70-85 years, ECOG performance status 0-1 versus 2 and in ³65 years and <70 years, ECOG performance status 2 versus 3.

* S-1 40mg/m2 orally twice daily on days 1 (evening) - 15 (morning)
* Capecitabine 1250mg/m2 orally twice daily on days 1 (evening) - 15 (morning) Treatment will be administered every 3 weeks and will be continued in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed gastric adenocarcinoma with recurrent or metastatic disease
2. Age of 70-85 years with Eastern Cooperative Oncology Group (ECOG) performance status 0-2 or age ≥65 and <70 with ECOG performance status ≥ 2
3. Measurable disease as defined by Response Evaluation Criteria In Solid Tumors (RECIST) Measurable lesions:

   * Lesions that can be accurately measured in at least one dimension by any of the following:

     * Computed tomography (CT) of abdomen, pelvis or thorax, if the longest diameter to be recorded is at least 10 mm with spiral CT
     * Chest x-ray, if the lung lesion to be recorded is clearly defined and surrounded by aerated lung and the diameter to be recorded is at least 20 mm- Physical examination, if the clinically detected lesions are superficial (e.g., skin nodule and palpable lymph nodes) and at least 10 mm
4. No prior chemotherapy for recurrent and/or metastatic disease (prior adjuvant/neoadjuvant chemotherapy is allowed at least 6 months has relapsed between completion of adjuvant/neoadjuvant therapy and enrolment into the therapy; prior S-1 or capecitabine is not allowed)
5. Adequate major organ function including the following:

   * Hematopoietic function:

     * absolute neutrophil count (ANC)≥1,500/mm3,
     * Platelet ≥ 100,000/mm3,
   * Hepatic function:

     * serum bilirubin =< 1.5 x upper limit of normal (ULN),
     * AST/ALT levels =< 2.5 x ULN ( 5 x ULN if liver metastases are present)
   * Renal function:

     * serum creatinine =< 1.5 x ULN
6. Patients should sign a written informed consent before study entry

Exclusion Criteria:

1. Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome (e.g. patients with partial or total gastrectomy can enter the study, but not those with a jejunostomy probe), or inability to take oral medication
2. Patients with active (significant or uncontrolled) gastrointestinal bleeding
3. Inadequate cardiovascular function:

   * New York Heart Association class III or IV heart disease
   * Unstable angina or myocardial infarction within the past 6 months
   * History of significant ventricular arrhythmia requiring medication with antiarrhythmics or significant conduction system abnormality
4. Serious concurrent infection or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy
5. Other malignancy within the past 3 years except non-melanomatous skin cancer or carcinoma in situ of the cervix
6. History of or current brain metastases
7. Psychiatric disorder that would preclude compliance
8. Known dihydropyrimidine dehydrogenase deficiency
9. Patients receiving a concomitant treatment with drugs interacting with S-1 or capecitabine such as flucytosine, phenytoin, warfarin, lamivudine, or allopurinol et al.
10. Patients with known active infection with HIV, HBV, or HCV
11. Major surgery within 4 weeks of start of study treatment, without complete recovery
12. Radiotherapy within 4 weeks of start of study treatment; 2 weeks interval allowed if palliative radiotherapy was given to bone metastatic site and patient recovered from any acute toxicity

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate each response rate of S-1 and capecitabine in the elderly and/or poor performance status patients with recurrent or metastatic gastric cancer | During Chemotherapy

SECONDARY OUTCOMES:
the duration of response, time to progression, progression-free survival,overall survival,the safety profiles,the quality of life,the CYP2A6 genetic polymorphism and its association with clinical outcomes in patients treated with S-1 | During study period

CONTACTS AND LOCATIONS:
Overall Officials: Sook Ryun Park, M.D, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea